CLINICAL TRIAL: NCT03798184
Title: Randomized Blind Clinical Trial, Four-armed Parallel of Clinical Performance of Prime&Bond Active in Self-etch or Selective-etch With or Without Bioglass
Brief Title: Clinical Performance of Prime&Bond Active in Self-etch or Selective-etch Mode With or Without Bioglass
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Cristina Pasarín Linares, Teaching Assistant, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2/2018
Record Dates: First submitted 2018-11-18; First posted 2019-01-09 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Self-etch; Selective-etch; Bioactive Glass; Direct Resin Composite Restoration; Non-carious Cervical Lesion; Universal Adhesive
Keywords: Prime&Bond Active; Bioactive glass; non-carious cervical lesion; direct resin composite

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Selective-etch with bioglass surface roughening (Experimental)
  Interventions: Procedure: Non-carious cervical lesion restoration
- Selective-etch without bioglass surface roughening (Active Comparator)
  Interventions: Procedure: Non-carious cervical lesion restoration
- Self-etch with bioglass surface roughening (Experimental)
  Interventions: Procedure: Non-carious cervical lesion restoration
- Self-etch without bioglass surface roughening (Active Comparator)
  Interventions: Procedure: Non-carious cervical lesion restoration

INTERVENTIONS:
Procedure: Non-carious cervical lesion restoration — Restoration of non-carious cervical lesions with Prime&Bond Active in self-etch or selective-etch mode with or without bioglass

SUMMARY:
Composite restoration of non-carious cervical lesions has always been a challenge for the clinician, considering that the most frequent cause of failure is retention loss.

Adhesion of composite restoration may be obtained by following four different etching techniques: total-etch in three steps, total-etch in two steps, self-etch in two steps, and self-etch in one step. Nowadays the tendency is to simplify the adhesive classic protocols. With the introduction of universal adhesives such as Prime&Bond Active (Dentsply Sirona) it is possible to obtain a total-etch pattern (enamel and dentine) without the classic etching technique with orthophosphoric acid.

On the other hand, there has been an increase in the awareness of the importance of remaining dental tissue preservation, avoiding preparation of a cavity. This is why it is now preferable to use bioactive glass in order to increase micromechanical retention on the dental surface, instead of the classical approach of preparing the surface with burs.

To date, there are no studies evaluating the clinical performance of the universal adhesive Prime&Bond Active on direct resin composite restoration of non-carious cervical lesions neither in a selective-etch mode (enamel etching) or a self-etch mode (no etching) or using sandblasting with bioactive glass. Therefore, the main objective of the study is to evaluate the retention rate of composite restorations using Prime&Bond Active and a previous sandblasted surface with bioglass in a three-year follow-up, as well as the presence of marginal discoloration, marginal integrity and marginal caries.

DETAILED DESCRIPTION:
The protocol to be followed in the study is as follows:

1. Obtention of a written informed consent of all participants.
2. Complete medical and dental clinical record.
3. Administration of anesthesia and absolute rubber dam isolation.
4. Cavity cleaning with a prophylactic brush and rubber cup with pumice.
5. Randomly assigning each non-carious cervical lesion to one of the four experimental groups:

   5.1. Selective enamel etching and surface roughening with bioglass 5.2. Selective enamel etching without surface roughening. 5.3. Self-etch and surface roughening with bioglass. 5.4. Self-etch without surface roughening.
6. In experimental groups which need surface roughening (group 5.1 and 5.3), sandblasting with bioactive glass will be used in enamel.
7. In experimental groups with selective enamel etch (5.1 and 5.2), 37 % orthophosphoric acid is applied for 15 seconds in enamel, followed by profuse washing with air/water spray for ten seconds and dried using air for 10 seconds without desiccating dentin.

   In groups 5.3 and 5.4 this step is omitted.
8. Application of universal adhesive Prime&Bond Active on enamel and dentin for 20 seconds. Subsequently, evaporation of the solvent is realized by applying air for 5 seconds and then light curing for 20 seconds.
9. Application of a "bulk fill" composite resin and light curing, following manufacturer's instructions.
10. Finishing and polishing of the restoration.
11. Monitoring and follow up: visits will be performed at six months, one year, two years and three years. In each evaluation, two independent clinicians who do not participate in the clinical procedures will evaluate each direct composite restoration according to USPHS criteria (Modified United States Public Health Service).

The primary objective is to evaluate the retention of the restoration. The secondary objectives are to evaluate marginal discoloration, marginal integrity and marginal caries.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years without systemic disease.
2. Presence of a non-carious cervical lesion with a minimum of 1.5 mm in depth and extent to dentin.
3. Non-carious cervical lesions in premolars and molars.

Exclusion Criteria:

1. Presence of rampant caries or advanced periodontal disease.
2. Consumption of > 2 cigarette pack/ day.
3. Presence of severe xerostomia or bruxism.
4. Methacrylate allergy.
5. Pregnancy.

Teeth with pulpal and/or periapical pathology, and endodontically treated teeth are excluded from the study.

Teeth with previous pulp capping or previous class V restorations will also be excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2018-11-19 (Actual); Primary Completion 2019-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Retention rate | Three years
  Presence of resin composite restorations of non-carious cervical lesions at the three-year follow-up examination.

SECONDARY OUTCOMES:
Marginal discoloration | Three years
  Presence of marginal staining between the restoration and tooth will be evaluated following USPHS criteria (Modified United States Public Health Service)
Marginal integrity | Three years
  The quality of the interface between restoration and tooth will be evaluated following USPHS criteria (Modified United States Public Health Service)
Marginal caries | Three years
  The presence of clinical diagnosis of caries will be evaluated following USPHS criteria (Modified United States Public Health Service)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Valencia, Valencia, Spain